CLINICAL TRIAL: NCT01087203
Title: A PHASE 2 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER, PARALLEL GROUP, PROOF OF CONCEPT STUDY OF THE ANALGESIC EFFECTS OF TANEZUMAB IN ADULT PATIENTS WITH DIABETIC PERIPHERAL NEUROPATHY
Brief Title: A Study Of The Analgesic (Pain-Relief) Effects Of Tanezumab In Adult Patients With Diabetic Peripheral Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091031; DPN PHASE 2B (Other: Alias Study Number)
Record Dates: First submitted 2010-03-11; First posted 2010-03-16 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: diabetic peripheral neuropathy; tanezumab; diabetic neuropathies; diabetic polyneuropathy; diabetic neuropathy painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tanezumab (Experimental)
  Interventions: Biological: Tanezumab
- Placebo (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Tanezumab — 20 mg subcutaneous injection every 8 weeks x 2 doses (at Baseline and week 8)
  Other Names: PF-04383119
  Arms: Tanezumab
Biological: placebo — Placebo to match tanezumab 20 mg subcutaneous injection every 8 weeks x 2 doses (at Baseline and week 8)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of the investigational drug, tanezumab, in adult patients with painful diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
This study was terminated on 18 November 2010 following a US FDA clinical hold for the tanezumab diabetic peripheral neuropathy clinical study which halted dosing and enrollment of patients on 19 July 2010 for potential safety issues.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus (high blood sugar) with HbA1c levels of ≤11% at Screening, and on a stable anti-diabetic medication regimen for the 30 days prior to randomization.
* Diagnosis of diabetic peripheral neuropathy pain in the legs or feet with decreased sensation in the feet or decreased/absent ankle jerk/ reflexes.
* Presence of ongoing pain due to diabetic peripheral neuropathy for at least 3 months.
* A pain score of greater than or equal to (≥) 4 for from diabetic peripheral neuropathy on the Numerical Rating Scale (NRS), a 11-point scale with 0 meaning no pain and 10 meaning worst pain at Screening.
* Be willing to stop all pain medications for diabetic peripheral neuropathy except for the limited use of acetaminophen (Tylenol) or ibuprofen-like (Motrin) medications between Screening and Baseline and not use prohibited pain medications throughout the duration of the study except as permitted by the study guidelines.

Exclusion Criteria:

* Painful neuropathies other than diabetic peripheral neuropathy.
* Other types of diabetic neuropathies.
* Patients with a past history of carpal tunnel syndrome (CTS) with signs or symptoms of CTS in the one year prior to Screening are not eligible for participation.
* Patients with fibromyalgia, regional pain caused by lumbar or cervical compression with radiculopathy or other moderate to severe pain.
* Patients with a present (current) history of sciatica are not eligible for participation.
* The presence of pain conditions that cannot be distinguished from diabetic peripheral neuropathy such as peripheral vascular disease.
* Amputations dues to diabetes.
* Patient with any clinically significant medical condition or laboratory abnormalities.
* History, diagnosis, or signs and symptoms of clinically significant neurological diseases (such as Alzheimer's disease, head trauma, epilepsy or stroke).
* History, diagnosis, or signs and symptoms of clinically significant psychiatric diseases (such as bipoar disorder or schizophrenia).
* History of known alcohol, analgesic or drug abuse within 2 years of Screening.
* Pregnant women, lactating mothers, women suspected of being pregnant, and women who wish to be pregnant during the course of clinical study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-03-30 (Actual); Primary Completion 2010-11-18 (Actual); Study Completion 2011-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (48):
- United States (48):
  - Alabama Orthopaedic Clinic, Mobile, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Dedicated Clinical Research, Goodyear, Arizona
  - Valley Radiology, Ltd., Goodyear, Arizona
  - Dedicated Clinical Research, Litchfield Park, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Anaheim Hills MRI Holdings, Inc, Anaheim Hills, California
  - Fullerton Neurology and Headache Center, Fullerton, California
  - NervePro Medical Corporation, Irvine, California
  - United Medical Imaging Healthcare (X-Ray Only), Irvine, California
  - Coordinated Clinical Research, La Jolla, California
  - LabCorp (Draw blood only), La Jolla, California
  - Alpine Clinical Research Center, Inc, Boulder, Colorado
  - JEM Research Institute, Atlantis, Florida
  - Medical Specialists of the Palm Beaches, Atlantis, Florida
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - SJS Clinical Research, Inc., Destin, Florida
  - White Wilson Medical Center, Fort Walton Beach, Florida
  - MD Clinical, Hallandale, Florida
  - Laszlo J. Mate, MD, North Palm Beach, Florida
  - Palm Beach Neurological Center, Advanced Research Consultants, Inc., Palm Beach Gardens, Florida
  - Neurology Clinical Research, Inc., Sunrise, Florida
  - Neurology Specialists of Decatur Research Center, Decatur, Georgia
  - Neurology Specialists of Decatur, Decatur, Georgia
  - Allied Physicians Inc d/b/a Fort Wayne Neurology, Fort Wayne, Indiana
  - American Health Network of IN, LLC, Greenfield, Indiana
  - Radiology Department, American Health Network, Greenfield, Indiana
  - Lee Research Institute, Lenexa, Kansas
  - Mid-Atlantic Medical Research Centers, Hollywood, Maryland
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Ozarks Community Hospital Christian County Clinic, Nixa, Missouri
  - Clinvest/A Division of Banyan Group, Inc., Springfield, Missouri
  - Montana Neuroscience Institute Foundation, Missoula, Montana
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - Joel Vandersluis, MD, Dayton, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Neurology and Neuroscience Center of Ohio, Toledo, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Mark A. Fisher M.D. -Private Practice, Oklahoma City, Oklahoma
  - Westmoreland Neurology Associates, Inc, Greensburg, Pennsylvania
  - The Neurology and Pain Clinic, Orangeburg, South Carolina
  - Centex Research/Pineloch Medical Center, Houston, Texas
  - Paragon Research Center, LLC, San Antonio, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Daniel B. Vine, MD, Salt Lake City, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - RGL Medical Services, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Bramson C, Herrmann DN, Carey W, Keller D, Brown MT, West CR, Verburg KM, Dyck PJ. Exploring the role of tanezumab as a novel treatment for the relief of neuropathic pain. Pain Med. 2015 Jun;16(6):1163-76. doi: 10.1111/pme.12677. Epub 2015 Jan 16. PMID 25594611
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091031&StudyName=A%20Study%20Of%20The%20Analgesic%20%28Pain-Relief%29%20Effects%20Of%20Tanezumab%20In%20Adult%20Patients%20With%20Diabetic%20Peripheral%20Neuropathy%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to tanezumab (RN624 or PF-04383119) subcutaneous injection on Day 1 and Week 8.
- Tanezumab: Tanezumab (RN624 or PF-04383119) 20 milligram (mg) subcutaneous injection on Day 1 and Week 8.
Period: Overall Study
Arm/Group | Placebo | Tanezumab
Started | 35 | 38
Completed | 3 | 3
Not Completed | 32 | 35
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Lack of Efficacy | 1 | 2
Not completed — Study terminated by sponsor | 27 | 27

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set included all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tanezumab | Total
Number analyzed (Participants) | 35 | 38 | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (11.6) | 61.6 (8.9) | 60.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 20 | 27 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Diabetic Peripheral Neuropathy (DPN) Pain Score at Week 16
Description: Participants assessed their DPN pain during the past 24 hours using 11-point Numeric Rating Scale (NRS) with score range of 0 (no pain) to 10 ( worst possible pain). Baseline score was calculated as the mean of the average pain scores over the 3 days in the initial pain assessment period. The Week 16 value was the average DPN Pain score calculated for the 7 days prior to and including Day 113 (Week 16).
Time Frame: Baseline, Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. Last Observation Carried Forward (LOCF) method of imputation was used.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 35 | 38
Units on a scale
  Baseline | 6.91 (1.50) | 6.59 (1.40)
  Change at Week 16 | -1.04 (1.92) | -2.10 (3.14)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab; Analysis of Covariance (ANCOVA) model with treatment as main effect, baseline value as covariate, and study site as a random effect was used; Test type: Superiority or Other; p = 0.025, ANCOVA; Least Squares (LS) mean difference = -1.22, 95% CI 2-sided [-2.28 to -0.16], Standard Error of Mean 0.53

2. Secondary Outcome: Change From Baseline in Average Diabetic Peripheral Neuropathy (DPN) Pain Score at Week 1, 2, 4, 6, 8, and 12
Description: Participant rated their DPN pain using 11-point NRS with score ranging from 0 (no pain) to 10 (worst possible pain) during past 24-hour period. Higher score indicated greater level of pain. Change: score at observation minus score at baseline.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. LOCF method of imputation was used.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 35 | 38
Units on a scale
  Baseline | 6.91 (1.50) | 6.59 (1.40)
  Change at Week 1 | -0.76 (1.31) | -0.97 (1.50)
  Change at Week 2 | -1.00 (1.67) | -1.31 (1.92)
  Change at Week 4 | -0.95 (1.75) | -1.78 (2.55)
  Change at Week 6 | -0.95 (1.68) | -2.04 (2.86)
  Change at Week 8 | -0.98 (1.83) | -2.16 (2.96)
  Change at Week 12 | -1.00 (1.89) | -2.14 (3.12)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab; Week 1: ANCOVA model with treatment as main effect, baseline value as covariate, and study site as a random effect was used; Test type: Superiority or Other; p = 0.332, ANCOVA; LS mean difference = -0.30, 95% CI 2-sided [-0.92 to 0.32], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: Placebo vs Tanezumab; Week 2: ANCOVA model with treatment as main effect, baseline value as covariate, and study site as a random effect was used; Test type: Superiority or Other; p = 0.297, ANCOVA; LS mean difference = -0.40, 95% CI 2-sided [-1.15 to 0.36], Standard Error of Mean 0.38
Statistical Analysis 3: Comparison: Placebo vs Tanezumab; Week 4: ANCOVA model with treatment as main effect, baseline value as covariate, and study site as a random effect was used; Test type: Superiority or Other; p = 0.029, ANCOVA; LS mean difference = -0.95, 95% CI 2-sided [-1.81 to -0.10], Standard Error of Mean 0.42
Statistical Analysis 4: Comparison: Placebo vs Tanezumab; Week 6: ANCOVA model with treatment as main effect, baseline value as covariate, and study site as a random effect was used; Test type: Superiority or Other; p = 0.010, ANCOVA; LS mean difference = -1.24, 95% CI 2-sided [-2.17 to -0.30], Standard Error of Mean 0.46
Statistical Analysis 5: Comparison: Placebo vs Tanezumab; Week 8: ANCOVA model with treatment as main effect, baseline value as covariate, and study site as a random effect was used; Test type: Superiority or Other; p = 0.009, ANCOVA; LS mean difference = -1.32, 95% CI 2-sided [-2.30 to -0.34], Standard Error of Mean 0.49
Statistical Analysis 6: Comparison: Placebo vs Tanezumab; Week 12: ANCOVA model with treatment as main effect, baseline value as covariate, and study site as a random effect was used; Test type: Superiority or Other; p = 0.015, ANCOVA; LS mean difference = -1.31, 95% CI 2-sided [-2.36 to -0.27], Standard Error of Mean 0.52

3. Secondary Outcome: Number of Participants With Cumulative Reduction From Baseline in Average Diabetic Peripheral Neuropathy (DPN) Pain Score at Week 16
Description: Participant rated their DPN pain using 11-point NRS with score ranging from 0 (no pain) to 10 (worst possible pain) during past 24-hour period. Higher score indicated greater level of pain.
Time Frame: Week 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 35 | 38
Participants
  Greater than (>) 0% | 23 | 24
  Greater than equal to (>=) 10% | 18 | 20
  >= 20% | 10 | 20
  >= 30% | 7 | 15
  >= 40% | 5 | 14
  >= 50% | 5 | 12
  >= 60% | 3 | 11
  >= 70% | 2 | 11
  >= 80% | 1 | 9
  >= 90% | 1 | 4
  = 100% | 1 | 4

4. Secondary Outcome: Number of Participants With at Least 30 Percent (%), 50%, 70% and 90% Reduction From Baseline in Average DPN Pain Score: Last Observation Carried Forward (LOCF)
Description: as for outcome 2
Time Frame: Week 1, 2, 4, 6, 8, 12, 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 35 | 38
Participants
  Week 1: >= 30% Reduction | 4 | 8
  Week 1: >= 50% Reduction | 2 | 3
  Week 1: >= 70% Reduction | 0 | 1
  Week 1: >= 90% Reduction | 0 | 0
  Week 2: >= 30% Reduction | 6 | 12
  Week 2: >= 50% Reduction | 3 | 7
  Week 2: >= 70% Reduction | 2 | 1
  Week 2: >= 90% Reduction | 1 | 0
  Week 4: >= 30% Reduction | 6 | 15
  Week 4: >= 50% Reduction | 3 | 9
  Week 4: >= 70% Reduction | 2 | 5
  Week 4: >= 90% Reduction | 1 | 1
  Week 6: >= 30% Reduction | 6 | 15
  Week 6: >= 50% Reduction | 2 | 10
  Week 6: >= 70% Reduction | 2 | 7
  Week 6: >= 90% Reduction | 1 | 3
  Week 8: >= 30% Reduction | 6 | 15
  Week 8: >= 50% Reduction | 4 | 12
  Week 8: >= 70% Reduction | 2 | 8
  Week 8: >= 90% Reduction | 1 | 5
  Week 12: >= 30% Reduction | 7 | 15
  Week 12: >= 50% Reduction | 4 | 12
  Week 12: >= 70% Reduction | 2 | 11
  Week 12: >= 90% Reduction | 1 | 4
  Week 16: >= 30% Reduction | 7 | 15
  Week 16: >= 50% Reduction | 5 | 12
  Week 16: >= 70% Reduction | 2 | 11
  Week 16: >= 90% Reduction | 1 | 4

5. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Worst and Average Pain Score at Week 8 and 16
Description: BPI-sf (Brief Pain Inventory-short form) is a participant-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during the 24-hour period prior to evaluation. It consists of 5 questions. Questions 1-4 measure the magnitude of pain at its worst and least (in the last 24 hours), average, and right now. Responses are provided by the participant on an 11-point numeric rating scale with anchors at 0 (No Pain) and 10 (Pain as bad as you can imagine). Question 5 consists of 7 item subsets (A to G) which measure the level of interference of pain on daily functions. Responses are given on an 11-point numeric rating scale with anchors at 0 (Does not interfere) and 10 (Completely interferes). The instrument is scored by item and by dimension, with lower scores indicating less pain or pain interference.
Time Frame: Baseline, Week 8, 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. LOCF method of imputation was used. Here, Overall Number of Participants Analyzed signifies participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 30 | 37
Units on a scale
  Worst Pain: Baseline | 7.33 (1.24) | 6.92 (1.38)
  Worst Pain: Change at Week 8 | -1.13 (1.70) | -2.38 (3.06)
  Worst Pain: Change at Week 16 | -1.10 (1.65) | -2.32 (3.06)
  Average Pain: Baseline | 6.17 (1.21) | 5.62 (1.40)
  Average Pain: Change at Week 8 | -0.77 (1.43) | -1.65 (2.14)
  Average Pain: Change at Week 16 | -0.73 (1.36) | -1.59 (2.15)

6. Secondary Outcome: Change From Baseline in Neuropathic Pain Symptom Inventory (NPSI) Total Score at Week 8 and 16: Last Observation Carried Forward (LOCF)
Description: Participant rated questionnaire to evaluate different symptoms of neuropathic pain (burning [superficial] spontaneous pain, pressing [deep] spontaneous pain, paroxysmal pain, evoked pain, and paresthesia/dyesthesia [P/D]) during past 24-hour period and included 10 descriptors quantified on a 0 (no symptoms) to 10 (worst symptoms imaginable) and 2 temporal items assessing duration of spontaneous ongoing and paroxysmal pain. Questionnaire generated a score in each of the relevant dimensions and a total score of 0-100. Higher score indicated a greater intensity of pain.
Time Frame: Baseline, Week 8, 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. Here, 'Overall Number of Participants Analyzed'= participants evaluable for this measure. 'Number Analyzed' = participants who were evaluable for this measure at given time point for each arm, respectively. LOCF method of imputation was used.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 30 | 36
Units on a scale
  Baseline | 0.50 (0.21) | 0.45 (0.18)
  Change at Week 8: number analyzed (Participants) | 23 | 31
  Change at Week 8 | -0.15 (0.21) | -0.20 (0.21)
  Change at Week 16: number analyzed (Participants) | 24 | 31
  Change at Week 16 | -0.13 (0.18) | -0.17 (0.22)

7. Secondary Outcome: Change From Baseline in BPI-sf Pain Interference Index and Pain Interference Score for General Activity, Walking Ability, Sleep and Normal Work at Week 8 and Week 16
Description: BPI-sf (Brief Pain Inventory-short form) is a participant-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during the 24-hour period prior to evaluation. It consisted of 5 questions. Questions 1-4 measure the magnitude of pain at its worst and least (in the last 24 hours), average, and right now. Responses were provided by the participant on an 11-point numeric rating scale with anchors at 0 (No Pain) and 10 (Pain as bad as you can imagine). Question 5 consisted of 7 item subsets (A to G) as being pain interference with general activity; mood; walking ability; normal work (outside home and housework); relations with other people; sleep and enjoyment of life. Responses were given on an 11-point numeric rating scale with anchors at 0 (Does not interfere) and 10 (Completely interferes). The instrument was scored by item and by dimension, with lower scores indicated less pain or pain interference.
Time Frame: Baseline, Week 8, 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. Here, 'Overall Number of Participants Analyzed= participants evaluable for this measure. 'Number Analyzed' =participants who were evaluable for this measure at given time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 30 | 37
Units on scale
  Pain Interference Index (PII);Baseline | 5.23 (2.36) | 4.71 (2.41)
  PII: Change at Week 8: number analyzed (Participants) | 23 | 32
  PII: Change at Week 8 | -1.12 (2.32) | -1.75 (3.15)
  PII: Change at Week 16: number analyzed (Participants) | 2 | 3
  PII: Change at Week 16 | -1.64 (0.51) | -1.24 (2.18)
  PI General Activity: Baseline | 5.30 (2.23) | 4.49 (3.02)
  PI General Activity: Change at Week 8: number analyzed (Participants) | 23 | 32
  PI General Activity: Change at Week 8 | -1.26 (2.20) | -1.81 (3.86)
  PI General Activity: Change at Week 16: number analyzed (Participants) | 2 | 3
  PI General Activity: Change at Week 16 | -2.00 (0.00) | -1.33 (3.51)
  PI Walking Ability: Baseline | 5.43 (2.50) | 5.54 (2.80)
  PI Walking Ability: Change at Week 8: number analyzed (Participants) | 23 | 32
  PI Walking Ability: Change at Week 8 | -1.09 (3.18) | -2.25 (3.21)
  PI Walking Ability: Change at Week 16: number analyzed (Participants) | 2 | 3
  PI Walking Ability: Change at Week 16 | -2.00 (1.41) | -2.33 (2.52)
  PI Sleep: Baseline | 5.70 (2.78) | 5.95 (2.59)
  PI Sleep: Change at Week 8: number analyzed (Participants) | 23 | 32
  PI Sleep: Change at Week 8 | -0.87 (2.69) | -2.34 (3.60)
  PI Sleep: Change at Week 16: number analyzed (Participants) | 2 | 3
  PI Sleep: Change at Week 16 | -1.00 (0.00) | -2.00 (1.00)
  PI Normal Work: Baseline | 5.33 (2.59) | 4.78 (2.89)
  PI Normal Work: Change at Week 8: number analyzed (Participants) | 23 | 32
  PI Normal Work: Change at Week 8 | -1.04 (2.53) | -1.44 (3.86)
  PI Normal Work: Change at Week 16: number analyzed (Participants) | 2 | 3
  PI Normal Work: Change at Week 16 | -1.50 (0.71) | -0.67 (3.51)

8. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Diabetic Peripheral Neuropathy (DPN) at Week 4, 8, 12 and 16
Description: The PGA is a global evaluation that utilizes a 5-point Likert scale with a score of 1 being the best (very good: Asymptomatic and no limitation of normal activities) and a score of 5 being the worst (very poor: Very severe symptoms which are intolerable and inability to carry out all normal activities).
Time Frame: Baseline, Week 4, 8, 12, 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. Here, 'Overall Number Analyzed' signifies those participants who were evaluable for this measure. LOCF method of imputation was used.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 30 | 37
Units on a scale
  Baseline | 3.17 (0.65) | 2.89 (0.61)
  Change at Week 4 | -0.47 (0.86) | -0.54 (0.84)
  Change at Week 8 | -0.63 (0.76) | -0.57 (0.93)
  Change at Week 12 | -0.63 (0.76) | -0.62 (0.89)
  Change at Week 16 | -0.63 (0.76) | -0.59 (0.90)

9. Secondary Outcome: Number of Participants With Improvement of at Least 2 Points in Patient's Global Assessment (PGA) of Diabetic Peripheral Neuropathy
Description: as for outcome 8
Time Frame: Week 4, 8, 12, 16
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 35 | 38
Participants
  Week 4 | 1 | 6
  Week 8 | 2 | 5
  Week 12 | 2 | 5
  Week 16 | 2 | 5

10. Secondary Outcome: Change From Baseline in Euro Quality of Life (EQ-5D)- Health State Profile Utility at Week 16
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression; 1 indicates better health state (no problems); 3 indicates worst health state (extreme problems). Scoring formula developed by Euro Quality of life group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicated a better health state.
Time Frame: Baseline, Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. 'Overall Number of Participants Analyzed'=participants evaluable for this measure. Here, 'Number Analyzed' signifies those participants who were evaluable for this measure at given time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 30 | 37
Units on a scale
  Baseline | 0.54 (0.29) | 0.62 (0.22)
  Change at Week 16: number analyzed (Participants) | 2 | 3
  Change at Week 16 | 0.00 (0.05) | -0.06 (0.11)

11. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Time Frame: Baseline up to Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 35 | 38
Days | 5.0 [5 to 5] | 21.0 [20 to 22]

12. Secondary Outcome: Number of Participants Who Used Rescue Medication
Description: Participants who did not experience adequate pain relief for DPN pain during the treatment period took acetaminophen 3000 mg/day up to 3 days/week as rescue medication.
Time Frame: Week 1, 2, 4, 6, 8, 12, 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. LOCF method of imputation was used. 'Overall Number of Participants Analyzed'=participants evaluable for this measure. Here, 'Number Analyzed' signifies those participants who were evaluable for this measure at given time point for each arm, respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 24 | 28
Participants
  Week 1: number analyzed (Participants) | 24 | 27
  Week 1 | 14 | 20
  Week 2 | 13 | 17
  Week 4 | 12 | 13
  Week 6 | 13 | 13
  Week 8 | 12 | 12
  Week 12 | 12 | 12
  Week 16 | 12 | 12

13. Secondary Outcome: Days Per Week of Rescue Medication Usage
Description: as for outcome 12
Time Frame: Week 1, 2, 4, 6, 8, 12, 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. LOCF method of imputation was used. Here, 'Overall Number of Participants Analyzed'=participants evaluable for this measure. 'Number Analyzed' signifies those participants who were evaluable for this measure at given time point for each arm, respectively.
Measure: Median (Full Range); unit: Days per week
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 24 | 28
Days per week
  Week 1: number analyzed (Participants) | 0 | 0
  Week 2 | 1 [0 to 7] | 1 [0 to 7]
  Week 4 | 1 [0 to 7] | 0 [0 to 7]
  Week 6: number analyzed (Participants) | 0 | 0
  Week 8 | 1 [0 to 7] | 0 [0 to 5]
  Week 12 | 1 [0 to 7] | 0 [0 to 5]
  Week 16 | 1 [0 to 7] | 0 [0 to 5]

14. Secondary Outcome: Amount of Rescue Medication Taken
Description: as for outcome 12
Time Frame: Week 1, 2, 4, 6, 8, 12, 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 24 | 28
mg/week
  Week 1: number analyzed (Participants) | 24 | 27
  Week 1 | 2666.67 (4090.46) | 2759.26 (3716.83)
  Week 2 | 2020.83 (2939.53) | 2178.57 (3174.59)
  Week 4 | 1354.17 (1997.17) | 1464.29 (2567.35)
  Week 6 | 1395.83 (1978.03) | 1250.00 (2420.97)
  Week 8 | 1354.17 (1997.17) | 1160.71 (2419.27)
  Week 12 | 1416.67 (2009.04) | 1160.71 (2419.27)
  Week 16 | 1416.67 (2009.04) | 1160.71 (2419.27)

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 112 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 112 days after last dose of study treatment (up to 169 days)
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 35 | 38
Participants
  AEs | 19 | 24
  SAEs | 0 | 1

16. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Values
Description: Criteria:Hemoglobin(Hgb),hematocrit,red blood cell(RBC)count:less than(<)0.8*lower limit of normal(LLN), mean cell Hgb,mean corpuscular volume,mean corpuscular Hgb concentration,mean platelet volume:<0.9*LLNor>1.1*upper limit of normal(ULN),platelet:<0.5*LLN >1.75* ULN, lymphocyte,neutrophil:<0.8*LLN or>1.2*ULN,basophil, eosinophil,monocyte:>1.2*ULN;bilirubin(total, direct,)>1.5*ULN, aspartate and alanine aminotransferase,alkaline phosphatase:> 3.0*ULN;gamma GT>3.0;cholestrol,triglycerides:>1.3*ULN; total protein, albumin:<0.8*LLN or>1.2*ULN ;blood urea nitrogen,creatinine:>1.3*ULN,uric acid>1.2*ULN;sodium <0.95*LLNor>1.05*ULN,potassium,chloride,calcium,bicarbonate, magnesium:<0.9*LLN or >1.1*ULN;phosphate<0.8*LLN or>1.2*ULN;glucose <0.6*LLNor>1.5*ULN,glycosylated Hgb>1.3*ULN,creatine kinase >2.0*ULN;urine(specific gravity<1.003or>1.030;pH <4.8or>8;glucose,ketone,proteins,blood/Hgb,bilirubin,nitrite>=1;WBC, RBC≥20/HPF;hyaline cast≥1;epithelial cell>=6;bacteria >1);serum pregnancy >=1.
Time Frame: Baseline up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. Here, 'Overall Number of Participants Analyzed'= total number of participants with at least one observation of the given laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 34 | 36
Participants | 33 | 32

17. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Following parameters were analyzed for ECG abnormality: PR interval, QRS interval, QT interval, QT interval corrected using the Fridericia's formula (QTcF), QT interval corrected using the Bazett's formula (QTcB), RR interval and heart rate (HR). Number of participants with clinically significant abnormal ECG findings reported as adverse events were presented.
Time Frame: Baseline up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 35 | 38
Participants | 1 | 4

18. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline Physical Examination
Description: Physical examination included examination of following sites in addition to general examination: abdomen, ears, extremities, eyes, head, heart, musculoskeletal, neck, nose, skin, throat, lungs and thyroid.
Time Frame: Baseline up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 35 | 38
Participants | 0 | 2

19. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Following parameters were analyzed for examination of vital signs: body temperature, blood pressure, pulse rate and respiratory rate. Number of participants with clinically significant abnormality in vital signs reported as adverse events were presented.
Time Frame: Baseline up to Week 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 35 | 38
Participants | 1 | 0

20. Secondary Outcome: Number of Participants With Anti Drug Antibody (ADA) for Tanezumab
Description: Human serum ADA samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semi-quantitative enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline, Week 8, 16, 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. Here, 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for Tanezumab 20 mg group.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab
Number analyzed (Participants) | 38
Participants
  Baseline | 0
  Week 8: number analyzed (Participants) | 32
  Week 8 | 0
  Week 16: number analyzed (Participants) | 31
  Week 16 | 1
  Week 24: number analyzed (Participants) | 3
  Week 24 | 0

21. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Weeks 2, 4, 8, 12, 16 and 24: Last Observation Carried Forward (LOCF)
Description: Neurologic examination assessed strength of groups of muscles of the head and neck, upper limbs and lower limbs, deep tendon reflexes and sensation (tactile, vibration, joint position sense and pin prick) of index fingers and great toes in order to complete the NIS. The NIS consists of 74 items (37 items assessed on the right side and 37 items assessed on the left side). Each item was rated on a scale of either 0 to 4 or 0 to 2 points, which were summed to calculate a total score. The NIS total score ranges from 0 to 244, where higher scores represent greater impairment.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16 and 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. 'Overall Number of Participants Analyzed'=participants evaluable for this measure. Here, 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group respectively. LOCF method of imputation was used.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 31 | 37
Units on a scale
  Baseline | 16.42 (10.42) | 15.86 (10.77)
  Change at Week 2: number analyzed (Participants) | 29 | 34
  Change at Week 2 | -1.90 (3.13) | -1.40 (4.93)
  Change at Week 4: number analyzed (Participants) | 30 | 36
  Change at Week 4 | -1.30 (4.02) | -0.35 (7.12)
  Change at Week 8: number analyzed (Participants) | 30 | 36
  Change at Week 8 | -1.63 (3.37) | -0.24 (5.40)
  Change at Week 12: number analyzed (Participants) | 30 | 36
  Change at Week 12 | -2.27 (3.87) | -1.19 (6.13)
  Change at Week 16: number analyzed (Participants) | 30 | 36
  Change at Week 16 | -1.58 (3.83) | -0.51 (6.31)
  Change at Week 24: number analyzed (Participants) | 30 | 36
  Change at Week 24 | -1.18 (3.77) | -0.51 (6.31)

22. Secondary Outcome: Change From Baseline Neuropathy Symptoms and Change (NSC) Score at Week 16: Last Observation Carried Forward (LOCF)
Description: The NSC (Neuropathy symptoms and change) is a standardized instrument and has been used to evaluate participants for number of symptoms of peripheral neuropathy. The NSC score included 38 (muscle weakness, Q1-19; sensation, Q20-29; and autonomic symptoms, Q30-38) symptom questions where the participants indicated experiencing the number of symptoms (to any severity). The score ranged from 0 to 38, with higher scores indicated more symptoms. The change score is the participant's comparison of the symptoms at last evaluation to the symptoms at onset. A change from baseline > 0 indicated increased neuropathy.
Time Frame: Baseline, Week 16
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 31 | 37
Units on a scale
  Baseline | 6.97 (4.04) | 7.57 (3.49)
  Change at Week 16: number analyzed (Participants) | 30 | 36
  Change at Week 16 | -1.07 (1.84) | -1.56 (2.85)

23. Secondary Outcome: Change From Baseline in Quantitative Sensory Testing (QST) at Week 16
Description: QST was performed on dorsum of foot and anterior thigh (at midpoint of a line from inguinal crease to midpoint of patella) to assess and quantify sensory function in lower extremity. Parameters were selected to assess small fiber function such as cooling detection threshold (mainly small diameter myelinated fibers, A delta), heat pain detection threshold (A delta and C fiber functions), and large fiber function via vibration detection threshold. normal deviate scores derived from a normal distribution of a reference population. A standard deviate score of 0 corresponds to 50th percentile of control population. Standard deviate score 1.96 corresponds to 95th percentile of normal distribution and -1.96 corresponds to 5th percentile of normal distribution. A normal deviate score indicated how many standard deviations higher (in case of positive normal deviate score) or lower (in case of negative normal deviate score) participant's value was relative to mean of reference population.
Time Frame: Baseline, Week 16
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. LOCF method of imputation was used. 'Overall Number of Participants Analyzed'=participants evaluable for this measure. Here, 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: Normal deviate score
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 30 | 38
Normal deviate score
  Baseline: VDT Left Foot: number analyzed (Participants) | 30 | 37
  Baseline: VDT Left Foot | 1.64 (1.14) | 1.47 (1.22)
  Baseline: CDT Left Foot: number analyzed (Participants) | 29 | 34
  Baseline: CDT Left Foot | 1.72 (0.87) | 1.54 (1.18)
  Baseline: HPDT 0.5 Left Foot: number analyzed (Participants) | 30 | 37
  Baseline: HPDT 0.5 Left Foot | 0.07 (1.88) | 0.38 (2.21)
  Baseline: HPDT 5.0 Left Foot: number analyzed (Participants) | 30 | 37
  Baseline: HPDT 5.0 Left Foot | 0.40 (2.23) | 1.06 (2.00)
  Baseline: HPDT 5.0-0.5 Left Foot: number analyzed (Participants) | 30 | 37
  Baseline: HPDT 5.0-0.5 Left Foot | 0.64 (1.39) | 0.80 (1.38)
  Baseline: VDT Left Thigh: number analyzed (Participants) | 29 | 38
  Baseline: VDT Left Thigh | 1.31 (1.16) | 1.07 (1.28)
  Baseline: CDT Left Thigh: number analyzed (Participants) | 28 | 38
  Baseline: CDT Left Thigh | 1.52 (1.09) | 1.76 (1.05)
  Baseline: HPDT 0.5 Left Thigh: number analyzed (Participants) | 30 | 35
  Baseline: HPDT 0.5 Left Thigh | -0.82 (1.50) | -0.48 (1.17)
  Baseline: HPDT 5.0 Left Thigh: number analyzed (Participants) | 30 | 35
  Baseline: HPDT 5.0 Left Thigh | -0.55 (1.70) | -0.04 (1.41)
  Baseline: HPDT 5.0-0.5 Left Thigh: number analyzed (Participants) | 30 | 35
  Baseline: HPDT 5.0-0.5 Left Thigh | 0.71 (1.32) | 0.71 (1.42)
  Change at Week 16: VDT Left Foot: number analyzed (Participants) | 30 | 37
  Change at Week 16: VDT Left Foot | -0.07 (0.66) | -0.01 (0.90)
  Change at Week 16: CDT Left Foot: number analyzed (Participants) | 29 | 34
  Change at Week 16: CDT Left Foot | 0.02 (0.50) | -0.16 (0.81)
  Change at Week 16: HPDT 0.5 Left Foot: number analyzed (Participants) | 30 | 37
  Change at Week 16: HPDT 0.5 Left Foot | -0.27 (1.52) | -0.04 (1.54)
  Change at Week 16: HPDT 5.0 Left Foot: number analyzed (Participants) | 30 | 37
  Change at Week 16: HPDT 5.0 Left Foot | 0.26 (1.53) | 0.09 (1.20)
  Change at Week 16:HPDT 5.0-0.5 Left Foot: number analyzed (Participants) | 30 | 37
  Change at Week 16:HPDT 5.0-0.5 Left Foot | 0.38 (1.27) | 0.21 (1.48)
  Change at Week 16: VDT Left Thigh: number analyzed (Participants) | 29 | 38
  Change at Week 16: VDT Left Thigh | -0.11 (0.88) | -0.06 (0.87)
  Change at Week 16: CDT Left Thigh: number analyzed (Participants) | 28 | 38
  Change at Week 16: CDT Left Thigh | 0.19 (0.95) | 0.09 (0.87)
  Change at Week 16: HPDT 0.5 Left Thigh: number analyzed (Participants) | 30 | 35
  Change at Week 16: HPDT 0.5 Left Thigh | -0.23 (1.36) | -0.27 (1.40)
  Change at Week 16: HPDT 5.0 Left: number analyzed (Participants) | 30 | 35
  Change at Week 16: HPDT 5.0 Left | -0.11 (1.26) | -0.05 (1.57)
  Change at Week 16:HPDT 5.0-0.5 Left Thigh: number analyzed (Participants) | 30 | 35
  Change at Week 16:HPDT 5.0-0.5 Left Thigh | 0.23 (1.57) | 0.22 (1.38)

24. Secondary Outcome: Change From Baseline in the Average Density of Protein Gene Product (PGP) 9.5-Positive Intraepidermal Nerve Fiber (IENF) at Week 16: LOCF
Description: IENF density was quantified in 3 millimeter (mm) immunostained skin punch biopsies containing epidermis and superficial dermis to evaluate the amount and morphological appearance of small diameter nerve fibers, both somatic and autonomic, in sensory neuropathies. IENF density was assessed from skin biopsies taken from the distal calves and distal thigh.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Fibers/mm
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 35 | 38
Fibers/mm
  Change at Week 16: Distal Calves | 0.40 (0.22) | -0.15 (0.21)
  Change at Week 16: Distal Thighs | 0.40 (0.45) | -0.30 (0.45)

25. Secondary Outcome: Plasma Tanezumab Concentration
Time Frame: Baseline(Day 1), Week 2, 4, 8, 12, 16, 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. Here, 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Tanezumab
Number analyzed (Participants) | 38
nanogram per milliliter (ng/mL)
  Day 1 | 13.66 (59.710)
  Week 2: number analyzed (Participants) | 33
  Week 2 | 1752 (610.54)
  Week 4: number analyzed (Participants) | 32
  Week 4 | 1316 (438.16)
  Week 8: number analyzed (Participants) | 33
  Week 8 | 591.9 (232.07)
  Week 12: number analyzed (Participants) | 29
  Week 12 | 475.9 (430.22)
  Week 16: number analyzed (Participants) | 32
  Week 16 | 265.6 (282.50)
  Week 24: number analyzed (Participants) | 3
  Week 24 | 97.77 (59.975)

26. Secondary Outcome: Serum Nerve Growth Factor (NGF)
Description: Serum samples were analyzed for determining total NGF concentration. Total NGF was analyzed using a validated, sensitive and specific immunoaffinity enrichment liquid chromatography tandem mass spectrometric (IA/LC/MS/MS) method.
Time Frame: Day 1, Week 8, 16, 24
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication. 'Overall Number of Participants Analyzed'=participants evaluable for this measure. Here, 'Number Analyzed' signifies those participants who were evaluable for this measure at given time points for each group respectively.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 32 | 37
picogram per milliliter (pg/mL)
  Day 1 | 48.10 (11.04) | 45.54 (12.25)
  Week 8: number analyzed (Participants) | 26 | 32
  Week 8 | 50.15 (11.21) | 4193.9 (1304)
  Week 16: number analyzed (Participants) | 27 | 32
  Week 16 | 46.12 (10.65) | 2811.3 (1284)
  Week 24: number analyzed (Participants) | 2 | 3
  Week 24 | 38.69 (4.47) | 2689.0 (316.8)

27. Other Pre Specified Outcome: Number of Participants With Subcutaneous Doses of Study Medication
Description: Number of participants are reported based on the maximum number of Subcutaneous doses of either tanezumab or placebo received.
Time Frame: Day 1 up to Week 8
Population: ITT analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tanezumab
Number analyzed (Participants) | 35 | 38
Participants
  1 dose | 32 | 35
  2 doses | 3 | 3

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Tanezumab
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/38
Other Adverse Events (participants affected / at risk) | 19/35 | 24/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=35) | Tanezumab (N=38)
Carotid Artery Stenosis (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=35) | Tanezumab (N=38)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Gravitational oedema (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
Irritability (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Areflexia (Nervous system disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 2
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hyporeflexia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Cataract operation (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Influenza (Infections and infestations) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated following a United States (US) Food and Drug Administration (FDA) partial clinical hold.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.